CLINICAL TRIAL: NCT07217821
Title: Stepped-Care Intervention of Music and Imagery to Assess Relief (SCIMITAR) Trial
Acronym: SCIMITAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Indiana Institute for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1903704-22-C-22; 66974 (Other: Henry Jackson Foundation)
Record Dates: First submitted 2025-10-15; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Musculoskeletal Pain; Veterans; Music Therapy
Keywords: chronic pain; veterans; musculoskeletal pain; music therapy; clinical trial
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: The SCIMITAR Trial is a 2-arm, parallel-group, randomized controlled trial. Participants will be randomized in a 1:1 allocation ratio to a stepped-care music intervention or a waitlist control.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to study arm allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped-care (Experimental): Step 1, Music Listening (ML): a music therapist will meet with the Veteran once to identify: musical tastes, preferences and activities. From this meeting a playlist will be compiled for the Veteran to listen to during the 4-week treatment period (step 1). Participants will be asked to listen to music for a minimum of 15 minutes per day at least 4 days per week.
  Step 2, Music Imagery (MI): Participants who move to step 2 will receive 8 weekly MI sessions over 8-10 weeks. The 8-session protocol has two stages. Stage 1 (sessions 1-4) is focused on learning to use music and imagery for self-regulation. Stage 2 (sessions 5-8) focuses on identifying and deepening inner resources and learning how to utilize them for self-care. Imagery is used during both stages, but becomes a central focus during Stage 2.
  Interventions: Behavioral: Stepped-care
- Waitlist control (No Intervention): Wait-list Control: Following the 6-month outcome assessment, participants in the wait-list control arm will be offered abbreviated treatment of 3 sessions with a music therapist (one session to introduce ML with the option to receive 2 additional MI sessions). Participants will also be offered a referral to music therapy services. Participants in the wait-list control arm (and stepped-care group) may receive other pain treatments such as analgesics and non-pharmacological options (e.g., physical therapy) for their chronic MSK pain. The wait-list control arm will provide an untreated comparison to stepped-care and music therapy to assess outcomes during the same trial period, while still offering participants music therapy at study end if desired.

INTERVENTIONS:
Behavioral: Stepped-care — Music listening in Step 1 and Music and imagery in step 2
  Other Names: Stepped-care music therapy
  Arms: Stepped-care

SUMMARY:
Th Stepped-Care Intervention of Music and Imagery to Assess Relief (SCIMITAR) Trial. SCIMITAR builds on our pilot study, the Feasibility and Acceptability of Music Imagery and Listening Interventions for Analgesia (FAMILIA), which demonstrated that telehealth delivery of music listening (ML) and music imagery (MI) interventions is feasible and acceptable to Veterans with chronic musculoskeletal pain. SCIMITAR leverages what we learned from FAMILIA into a fully powered trial, harnessing the benefits of sequential ML and MI into a stepped-care, music therapy intervention via telehealth for Veterans needing relief from pain.

DETAILED DESCRIPTION:
More than 100 million Americans have chronic pain. Chronic pain affects 40%-70% of Veterans and is a leading cause of disability, with a substantial negative impact on millions of veterans' lives. Chronic pain is frequently accompanied by psychological comorbidity that adds to patient suffering and complicates treatment. Veterans with pain and PTSD demonstrate greater pain, depression, and healthcare utilization, and patients with comorbid pain and depression have worse outcomes than patients with pain or depression alone. Musculoskeletal (MSK) pain conditions are widespread, accounting for two-thirds of all clinical visits for pain. There is a pressing need to provide effective, non-pharmacological treatment to Veterans with chronic MSK pain. To improve pain-related outcomes, the VA recommends an integrative and stepped-care approach to pain management, including non-pharmacological treatments.

The SCIMITAR Trial is a 2-arm, parallel group, randomized controlled trial. After providing informed consent and completing their baseline assessment, participants will be randomized in a 1:1 allocation ratio to a stepped-care music intervention or waitlist control. The study population will include 180 Veterans with chronic MSK pain.

ELIGIBILITY:
Inclusion Criteria:

* musculoskeletal pain in the low back, cervical spine, or extremities (hips, knees, or shoulders) for ≥ 3 months
* at least moderate pain severity, defined as a PEG score ≥ 4 on a 0 (no pain) to 10 (worst pain)
* access to computer, tablet, or smartphone
* ability to pass a technology assessment

Exclusion Criteria:

* Past month hospitalization for medical or psychiatric illness
* housing insecurity
* suicidal ideation with current intent/plan
* hearing or cognitive impairment that may interfere with music listening or abstract thinking needed for imagery work
* currently receiving music therapy services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Pain Interference | baseline, 1, 3, and 6 months
  Assesses how pain interferes with 7 activities of daily living

SECONDARY OUTCOMES:
Numeric rating scale | baseline, 1, 3, and 6 months
  Assess pain severity
Patient Global Impression of Change | 1, 3, and 6 months
  Assess treatment response
PROMIS Sleep Scale | baseline, 1, 3, and 6 months
  Assesses quality of sleep
GAD-7 Anxiety | baseline, 1, 3, and 6 months
  Assesses anxiety symptoms
PHQ-9 Depression | baseline, 1, 3, and 6 months
  Assesses depression symptoms
PC PTSD Screen | baseline, 1, 3, and 6 months
  Screens for PTSD
Perceived Stress Scale | baseline, 1, 3, and 6 months
  Assesses stress
Mood regulation (B-MMR) | baseline, 1, 3, and 6 months
  Assesses ability to regulate mood

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Health Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss with potential collaborators on a case-by-case basis.